CLINICAL TRIAL: NCT05859958
Title: ABO Blood Group Type Association With COVID-19 Severity - A Single Center Study
Brief Title: ABO Blood Group Type Association With COVID-19 Severity
Status: Completed | Type: Observational
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-53
Record Dates: First submitted 2023-05-15; First posted 2023-05-16 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Blood Group Antigen Abnormality; Blood Group Incompatibilities; Diabetes Mellitus; COVID-19 Pandemic
MeSH Terms: conditions — COVID-19; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABO + Group: All patient with blood type that does not include Rhesus Factor and COVID-19 Diagnosis
  Interventions: Other: No Intervention
- ABO - Group: All patient with blood type that does not include Rhesus Factor and COVID-19 Diagnosis
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Difference in outcomes in patients with COVID-19 diagnosis and ABO blood groups

SUMMARY:
The COVID-19 pandemic has caused a significant healthcare burden and remains a heavily researched disease entity. Originating in Wuhan, China in late 2019, SARS-CoV-2 has infected over 600 million individuals worldwide. ABO blood groups have been known to increase the human body's susceptibility to different pathogens, such as hepatitis B virus, MERS-COV, SARS-COV, norovirus, and malaria, to name a few. As such, the association of ABO blood groups and COVID-19 infection and disease severity has come into question.

DETAILED DESCRIPTION:
The COVID-19 pandemic has caused a significant healthcare burden and remains a heavily researched disease entity. Originating in Wuhan, China in late 2019, SARS-CoV-2 has infected over 600 million individuals worldwide. ABO blood groups have been known to increase the human body's susceptibility to different pathogens, such as hepatitis B virus, MERS-COV, SARS-COV, norovirus, and malaria, to name a few. As such, the association of ABO blood groups and COVID-19 infection and disease severity has come into question.

Early reports have indicated a significant relationship of ABO blood group types to the risk of infection with SARS-CoV-2. Specifically, the first systematic review and meta-analysis by Wu et al. in October 2020 cited that blood type A had increased risk for infection with SARS-CoV-2 and blood type O had decreased risk of infection. Another early meta-analysis by Zaidi et al. cited that blood type A had increased odds of infection, type O had decreased odds of infection, type AB had increased risk of disease severity, and type B had decreased risk of demise.

As more multi-national data became available, as a result of global concerted efforts, larger studies produced data to further investigate this connection. Overall, the majority of studies reproduced similar data: type O had decreased risk of infection with SARS-CoV-2, while type A had increased risk of infection. One study in the United Kingdom failed to produce a relationship between blood types and COVID-19. As more data became available, several studies were able to study the association of blood group type with mortality and disease severity; however, the data regarding this is inconsistent. Gutierrez-Valencia et al. did not find an association with blood types and ICU admission or mechanical ventilation; however, they did note an increased risk of mortality in blood type A. Liu et al. and Pereira et al. demonstrated that there is also increased risk of mortality in blood type A. Jerico et al. noted a lower risk for ICU admission in blood type O. Goel et al. noted an increased risk of disease severity in blood type A. As evident, it seems that blood type A has increased risk of mortality and, likely, disease severity.

In this study, we aim to evaluate association of blood types with mortality and disease severity at a county hospital in Southern California. We will review charts for patients infected with SARS-CoV-2 during a two-year time period, evaluating mortality, oxygen requirements, and patient historical factors. Through this study, we aim to gain a better understanding of how blood group types may affect patient outcomes in the setting of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* COVID-19 confirmed by laboratory testing (ICD10 U07.1)
* Pneumonia due to COVID-19 (ICD10 J12.82)
* Multisystem inflammatory syndrome from COVID in adults (ICD10 M35.81)
* Adult respiratory distress syndrome (ICD10 J80)
* Abnormal pulmonary function test (ICD10 R94.2)
* Intensive care unit admission for COVID-19

Exclusion Criteria:

* COVID-19 Diagnosis under 18 years of age
* COVID in pregnancy (O98.52, O98.511, O98.512, O98.513, O98.519, O98.53)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To evaluate blood types and their associations with COVID-19 disease severity in patients older than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Length of total hospital stay from admission in the hospital is defined as the time frame between admission and discharge. The time frame of collection until the event occurred was 360 days.
  The time spent hospitalized in days.
Hospital Mortality | 28 days
  Survival within the first 28 days
Discharge disposition | 360 days
  Location of discharge after hospital course completed

CONTACTS AND LOCATIONS:
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu BB, Gu DZ, Yu JN, Yang J, Shen WQ. Association between ABO blood groups and COVID-19 infection, severity and demise: A systematic review and meta-analysis. Infect Genet Evol. 2020 Oct;84:104485. doi: 10.1016/j.meegid.2020.104485. Epub 2020 Jul 30. PMID 32739464
- [Background] Zaidi FZ, Zaidi ARZ, Abdullah SM, Zaidi SZA. COVID-19 and the ABO blood group connection. Transfus Apher Sci. 2020 Oct;59(5):102838. doi: 10.1016/j.transci.2020.102838. Epub 2020 Jun 3. No abstract available. PMID 32513613
- [Background] Gutierrez-Valencia M, Leache L, Librero J, Jerico C, Enguita German M, Garcia-Erce JA. ABO blood group and risk of COVID-19 infection and complications: A systematic review and meta-analysis. Transfusion. 2022 Feb;62(2):493-505. doi: 10.1111/trf.16748. Epub 2021 Nov 19. No abstract available. PMID 34773411
- [Result] Fan Q, Zhang W, Li B, Li DJ, Zhang J, Zhao F. Association Between ABO Blood Group System and COVID-19 Susceptibility in Wuhan. Front Cell Infect Microbiol. 2020 Jul 21;10:404. doi: 10.3389/fcimb.2020.00404. eCollection 2020. PMID 32793517